CLINICAL TRIAL: NCT04539028
Title: Emergency General Surgery for Non-trauma - A Prospective Observational Study
Brief Title: Emergency General Surgery for Non-trauma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Rifat Latifi, Chairman, Department of Surgery, New York Medical College
Other Study IDs: 12811
Record Dates: First submitted 2019-07-31; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Bowel Obstruction
Keywords: Emergency Abdominal surgery, Acute abdomen
MeSH Terms: conditions — Intestinal Obstruction; Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Emergency Abdominal surgery — Emergency Abdominal surgery

SUMMARY:
This study will observe the postoperative morbidity and mortality trends in patients with non- traumatic abdominal pathology who will undergo emergency general surgery. This prospective study will help us in establishing a prospective de-identified registry that may be used to further research this cohort in the future.

DETAILED DESCRIPTION:
Primary Objectives The first objective of this study is to analyze postoperative outcomes as well as morbidity and mortality trends for this sick cohort of patients with non- traumatic abdominal pathology who will undergo emergency general surgery. The second objective of this study is to establish a prospective de-identified registry database that may be used to further study this cohort in the future.

CHARACTERISTICS OF THE STUDY POPULATION

1. Target Population The target population will be all patients between the ages of 18-99, regardless of sex, racial or ethnic background that underwent emergent laparotomy and planned/unplanned re-laparotomy. Variables to be analyzed in the study are in the attached data collection excel sheet.
2. Key Inclusion Criteria

   * All adult patients ages 18-99, regardless of sex, racial or ethnic background who will undergo or underwent emergency abdominal surgery for acute abdomen due to perforated viscus, acute bowel obstruction, bowel ischemia, acute or gangrenous gall bladder, post-operative complications such as anastomotic leaks after bowel anastomosis, abdominal compartment syndrome,enterocutaneous/enteroatmospheric fistula or bleeding.
   * Investigators will also include patients after organ transplant that will undergo emergent surgery for post-operative bleeding, anastomotic leak or organ ischemia.
   * As well as any patients undergoing bariatric surgery or colorectal procedures that develop any complication that might need return to the operating room emergently will also be included in the study from 2019 at Westchester Medical Center.
3. Key Exclusion Criteria

   * Elective delayed repair for surgery done after clinic follow-up.
   * Age < 18 years or greater than 89 years of age
4. Vulnerable Populations Vulnerable populations such as children, fetuses, neonates, or prisoners will not be included in this research study.
5. Study Design This study is a prospective observational study of patients that are admitted to Westchester Medical Center and undergo emergency general surgery. Each chart will be reviewed for pre-op, intra-op, and post-op variables outlined in data collection tool. Data will be collected until one year after discharge on follow up visits. At the end of the study, all of this data will be analyzed to determine if there are any trends in mortality or morbidity for these patients. The variables will then be compared by using step-wise logistic regression techniques.
6. Study Duration The study will take place between 02/10/2019 to 1/31/2022.
7. Number of Subjects The study team/Investigators aim to enroll approximately 300 subjects.

Follow up:

Study team will follow patients for 1 year after discharge and the follow up visits are conducted in the clinic after 30 days, 3 months, 6 months and 1 year of discharge. Investigators will examine incision sites, drains if present and enquire about adequacy of pain control and unplanned readmission including any therapeutic or diagnostic procedures done, number of hospital days during readmission.

Statistical Analysis Chi-square difference tests will be used to assess significant differences in predictors on categorical outcomes. T-tests will be used to assess mean differences in predictors on continuous outcomes. Univariable and multivariable logistic regression analyses will be conducted for outcomes such as all-cause mortality, pneumonia, sepsis, and multi-organ failure. Univariable and multivariable linear regression will be performed for hospital length of stay.

Confidentiality Subjects will be recruited, consented, and data from medical record data will be gathered prospectively. Data will be obtained on a patient's pre and perioperative details, their interventions, and final outcomes. Two data files will be maintained: a master file and an analysis (de-identified data) file.

1. Master File: Identifiable Data: Medical Record Numbers, date of birth, admission date, discharge date, ICU admission date and time, any readmission data collected during follow-up, and date of death (if applicable) will be collected as part of this study and stored electronically in an Excel file (Master List). Each subject will be assigned an ID ( 3 digit number) under which all the collected information will be stored for that subject. This file will be password-protected. The Master File will also contain a unique id that is used to link identifiable data with the de-identified dataset used for analysis.
2. The de-identified dataset will also be password protected and each record will be organized by the unique ID. This file will include derived fields such as length of stay that will be calculated using data stored in the Master File.

RISK/BENEFIT ASSESSMENT

1. Potential Study Risks This study involves no more than minimal risk to subjects as it involves no additional treatment/interventions. There is the potential risk for breach of confidentiality. However, all research personnel will be trained in how to maintain confidentiality and protect PHI. Only research staff will have access to the de-identified information. Hard copies are locked in a file cabinet and electronic files are saved in password protected computers issued by WMC and computer access will be monitored.
2. Potential Study Benefits There are no direct benefits to the subjects participating in this study. Future patients may benefit from the information obtained from this prospective observational study. For example, to date, no large-scale prospective study on damage control surgery in trauma and non-traumatic pathology has been identified. If investigators observe an association between the variable that affects morbidity or mortality, investigators may be able to initiate appropriate therapy in a more timely fashion for future patients.
3. Data and Safety Monitoring Data Safety and monitoring will be done by the Principal Investigator and the research team. Data will be queried from the database and kept in a password protected excel spreadsheet. Only the PI will have the access to the data which has been coded with the subject identifier. The PI designated research team members will have the access to the de-identified data. Data will be stored on secure password protected Westchester Medical Center (WMC) servers. The only hard copies of patient documents will be the consent forms and HIPAA forms, which will be stored in a study binder that will be kept in locked cabinets in the PI's office. The identifiable PHI will be destroyed as soon as the data analysis is complete. The de-identified PHI will be kept in a database for future research. The hard copies of the study documents will be shredded.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients ages 18-99, regardless of sex, racial or ethnic background who will undergo or underwent emergency abdominal surgery for acute abdomen due to perforated viscus, acute bowel obstruction, bowel ischemia, acute or gangrenous gall bladder, post-operative complications such as anastomotic leaks after bowel anastomosis,abdominal compartment syndrome,enterocutaneous/enteroatmospheric fistula or bleeding.
* Investigators will also include patients after organ transplant that will undergo emergent surgery for post-operative bleeding, anastomotic leak or organ ischemia.
* As well as any patients undergoing bariatric surgery or colorectal procedures that develop any complication that might need return to the operating room emergently will also be included in the study from 2019 at Westchester Medical Center.

  3. Key Exclusion Criteria
* Elective delayed repair for surgery done after clinic follow-up.
* Age < 18 years or greater than 89 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients ages 18-99, regardless of sex, racial or ethnic background who will undergo or underwent emergency abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
morbidity and mortality | 1 year
  The objective of this study is to analyze postoperative outcomes as well as morbidity and mortality trends for this sick cohort of patients with non- traumatic abdominal pathology who will undergo emergency general surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rifat Latifi, MD, Principal Investigator — Chairman, Department of Surgery
Locations (1):
- Westchester Medical Center, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No